CLINICAL TRIAL: NCT04612699
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study of Jaktinib in Patients With Moderate-to-Severe Plaque Psoriasis
Brief Title: A Phase 2 Study of Jaktinib in Participants With Moderate to Severe Psoriasis
Acronym: PSO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZGJAK010
Record Dates: First submitted 2020-10-29; First posted 2020-11-03 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Moderate-to-Severe Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Jaktinib 50mg Bid (Experimental): Jaktinib 50mg Bid+ Placebo 50mg Bid+ Placebo 75mg Bid
  Interventions: Drug: Jaktinib; Drug: Placebo
- Jaktinib 75mg Bid (Experimental): Jaktinib 75mg Bid+ Placebo 50mg*2 Bid
  Interventions: Drug: Jaktinib; Drug: Placebo
- Jaktinib 100mg Bid (Experimental): Jaktinib 50mg*2 Bid+ Placebo 75mg Bid
  Interventions: Drug: Jaktinib; Drug: Placebo
- Placebo (Placebo Comparator): Placebo 50mg*2 Bid+ Placebo 75mg Bid
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Jaktinib — Administered orally
  Arms: Jaktinib 100mg Bid; Jaktinib 50mg Bid; Jaktinib 75mg Bid
Drug: Placebo — Administered orally

SUMMARY:
This is study designed to investigate the efficacy and safety of Jaktinib in the treatment of participants with moderate to severe, chronic plaque psoriasis as assessed by the Psoriasis Area and Severity Index (PASI) score and routine safety assessments.

ELIGIBILITY:
Inclusion Criteria:

* 18~65 years old (including lower limit), no gender limit；
* You must have active chronic plaque psoriasis for at least 6 months prior to entry into the study；
* You must have active plaque psoriasis covering at least 10% body surface area； You must have Psoriasis Area and Severity Index (PASI) score of at least 12；You must have Static Physician's Global Assessment (sPGA) score of at least 3；
* The patient can communicate well with the investigator and follow the research and follow-up procedures；
* Understand and voluntarily sign the informed consent form.

Exclusion Criteria:

* You must not have prior treatment with an oral Janus kinase (JAK) inhibitor；
* You must not have received a phototherapy within 4 weeks prior to entry into the study；
* You must not have a history of active hepatitis B, hepatitis C, or human immunodeficiency virus (HIV)；
* You must not have a history of chronic alcohol abuse or intravenous (IV) drug abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Psoriasis Area and Severity Index Score ≥75% (PASI 75) Improvement (Efficacy of Jaktinib in Participants With Moderate to Severe Plaque Psoriasis. Measure: Psoriasis Area and Severity Index [PASI]) | Week 12
  The PASI combines assessments of the extent of body-surface involvement in 4 anatomical regions (head, trunk, arms, and legs) and the severity of desquamation (scaling), erythema (redness), and plaque induration/infiltration (thickness) in each region, yielding an overall score of 0 for no psoriasis to 72 for the most severe disease.

SECONDARY OUTCOMES:
Percentage of Participants Achieving a Static Physician Global Assessment (sPGA) of (0, 1) (Efficacy of Jaktinib in Participants With Moderate to Severe Plaque Psoriasis. Measure: Static Physician Global Assessment [sPGA]) | Week 8、12、16、20、24
  The sPGA is a physician's determination of the participant's psoriasis lesions overall at a given time point categorized by descriptions for induration, erythema, and scaling. For the analysis of responses, the participant's psoriasis is assessed as clear

CONTACTS AND LOCATIONS:
Overall Officials: Xinghua Gao, PhD, Principal Investigator — First Hospital of China Medical University
Locations (1):
- The First Affiliated Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No